CLINICAL TRIAL: NCT04813185
Title: Preventing Retaliatory Gun Violence in Violently Injured Adults: A RCT of a Hospital-Based Intervention
Brief Title: Preventing Retaliatory Gun Violence in Violently Injured Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20020621; R01CE003296 (NIH)
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Violence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Adults who will not receive BTG services and will receive treatment as usual (TAU) in the hospital.
- In-hospital intervention (Experimental): Adults randomized to Bridging the Gap (BTG) services will receive a hospital-based violence prevention program with 6-months of community case management and a firearm counseling program.
  Interventions: Behavioral: Bridging the Gap

INTERVENTIONS:
Behavioral: Bridging the Gap — Bridging the Gap Bridging the Gap is a hybrid model for violence prevention which integrates a hospital-based brief violence intervention (BVI) delivered to the patient while in hospital with a wrap-around community case management prevention strategy.
  Firearm Counseling Program The firearm counseling program was developed to be administered in the hospital alongside the 6-step intervention program, as well as in the patient's home after hospital discharge. The firearm safety counseling program includes 3 components aimed at understanding patient risk, reducing firearm-related violence risk-factors, and helping patients increase firearm safety practices.
  Arms: In-hospital intervention

SUMMARY:
The purpose of this research study is to find out if a hospital-based violence intervention (Bridging the Gap) is effective for reducing violence. The researchers think that adults who receive Bridging the Gap will see greater improvements than those who do not receive the intervention. This study will allow them to learn more about the intervention's effectiveness. The study will also help them understand if the violence intervention affects other behaviors, such as firearm use, drug use, aggression, risky behaviors, and rates of violent re-injury.

DETAILED DESCRIPTION:
Approximately 616 patients will enroll in this study. Participants will be asked to complete sessions about behavior, personality, and experiences. Participants will be randomized into a study group (either Bridging the Gap or Treatment as Usual) by drawing a number. If patients agree to the study but do not like the group they are assigned to, they can request to switch groups. Participants assigned to the Treatment as Usual intervention will receive a brief violence awareness brochure during your hospital stay. Participants assigned to the Bridging the Gap intervention will receive an in-hospital intervention and, once released from the hospital, will receive 6-months of community case management services. The study team thinks that adults who receive the Bridging the Gap intervention will see greater improvements than adults who do not receive the intervention. This study will allow them to learn more about the intervention's effectiveness.

During these study sessions participants will complete questionnaires about exposure to traumatic events, symptoms of trauma, history of suicide, aggression and violence, antisocial personality traits, illegal behaviors, substance use, and mental health. Participants will complete several tasks which measure cognitive ability, such as problem-solving, attention/concentration, and decision-making. They will also complete a clinical interview that covers antisocial personality traits and behaviors, including history of aggressive behavior and substance use. These interviews will be video recorded. These recordings will be used to help score the interviews and for training purposes. Information will also be collected from participant's medical records, including demographic information, history and reason for past hospitalizations, mental health history, and substance use reports, as well as a criminal background check.

The surveys take about 2 hours to complete. Participants will complete these questionnaires again 6 and 12 months later. Participation in this study will last up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* They receive treatment in the hospital for a violence-related injury (e.g., gunshot wound)
* They are 18 years or older
* They are English speaking
* They are eligible for BTG services (which includes living within the BTG catchment area for the hospital; Richmond City and neighboring counties)

Exclusion Criteria:

* Non-English speaking
* Age <18
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Firearm-related violence | 12-months
  Number of firearm-related violence incidents will be measured multiple ways including self-report and a semi-structured clinical assessment of non-convicted firearm-related violence. Incidents will be summed to yield a single count of unique firearm-related violence incidents for each participant.
Firearm-related re-injury | 12-months
  Number of firearm-related re-injury incidents will be measured multiple ways including self-report and hospital records. Incidents will be summed to yield a single count of unique firearm-related re-injuries for each participant.
Firearm-related mortality | 12-months
  Collected from hospital records and National Death Index

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomson, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No